CLINICAL TRIAL: NCT00298350
Title: Phase 2 Study of the Treatment of Antiretroviral Treatment-Experienced Subjects Comparing Ritonavir-Boosted GS-9137 (GS-9137/r) vs. a Comparator Ritonavir-Boosted Protease Inhibitor (CPI/r) in Combination With Background ART.
Brief Title: Ritonavir-Boosted GS-9137 vs. Ritonavir-Boosted Protease Inhibitor(s) in Combination With Background ART.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Kitty Yale, Gilead Sciences INC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-183-0105
Record Dates: First submitted 2006-02-28; First posted 2006-03-02 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 2008-07

CONDITIONS: HIV; HIV-1; Human Immunodeficiency Virus
Keywords: Phase 2; Phase II; Randomized; Controlled; Comparator; Partially Blind; Protease Inhibitors; Integrase Inhibitors; Antiviral Agents; Antiretroviral Agents; ART; ARV; Highly Activity Antiretroviral Therapy; HAART; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: GS-9137 - A Novel HIV-1 Integrase Inhibitor

SUMMARY:
The purpose of this study is to evaluate the non-inferiority of ritonavir-boosted GS-9137 relative to a ritonavir-boosted Comparator Protease Inhibitor when used as part of combination antiretroviral regimens in subjects who have failed, or are failing, protease inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* HIV RNA greater than or equal to 1000 c/mL.
* Failed/Failing protease inhibitor based antiretroviral therapy.
* Stable antiretroviral therapy for greater than or equal to 30 days prior to screening.
* Negative Serum Pregnancy Test.
* GFR by Cockcroft Gault greater than or equal to 80 mL/min.
* AST & ALT less than or equal to 2.5x ULN.
* Total Bilirubin less than or equal to 1.5 mg/dL.
* Albumin greater than 3.5 mg/dL.
* Prothrombin Time INR 1.0-1.4
* Platelets greater than or equal to 50,000.
* Hemoglobin greater than or equal to 8.0 mg/dL.
* Absolute Neutrophil Count greater than or equal to 1000.

Exclusion Criteria:

* New AIDS defining condition within 30 days of baseline.
* Prior treatment with HIV-1 integrase inhibitor (except patients from 183-101).
* Ascites or encephalopathy.
* Breast Feeding.
* Cancer Diagnosis (besides Kaposi Sarcoma or Basal Cell Carcinoma).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2006-02; Primary Completion 2007-06 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (54):
- United States (52):
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Beverly Hills, California
  - Fountain Valley, California
  - Long Beach, California
  - Los Angeles, California
  - Newport Beach, California
  - Oakland, California
  - San Diego, California
  - San Francisco, California
  - Stanford, California
  - Sunnyvale, California
  - Torrance, California
  - Denver, Colorado
  - Norwalk, Connecticut
  - Washington D.C., District of Columbia
  - Atlantis, Florida
  - Fort Lauderdale, Florida
  - Miami, Florida
  - North Miami Beach, Florida
  - North Palm Beach, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Decatur, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Detroit, Michigan
  - St Louis, Missouri
  - Henderson, Nevada
  - Hillsborough, New Jersey
  - Santa Fe, New Mexico
  - Albany, New York
  - Manhasset, New York
  - New York, New York
  - Huntersville, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - Annandale, Virginia
  - Hampton, Virginia
  - Seattle, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
- Puerto Rico (2):
  - San Juan
  - Santurce

REFERENCES:
- [Derived] Zolopa AR, Berger DS, Lampiris H, Zhong L, Chuck SL, Enejosa JV, Kearney BP, Cheng AK. Activity of elvitegravir, a once-daily integrase inhibitor, against resistant HIV Type 1: results of a phase 2, randomized, controlled, dose-ranging clinical trial. J Infect Dis. 2010 Mar 15;201(6):814-22. doi: 10.1086/650698. PMID 20146631
- See also: Gilead Website — http://www.Gilead.com